CLINICAL TRIAL: NCT01905670
Title: Multicenter, Prospective Evaluation of Safety and Performance of the WiCS-LV System in Patients Indicated for Cardiac Resynchronization Therapy
Brief Title: Safety and Performance of Electrodes Implanted in the Left Ventricle
Acronym: SELECT-LV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EBR Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EBR-02494; CIV-13-04-010803 (Other: EUDAMED)
Record Dates: First submitted 2013-07-19; First posted 2013-07-23 (Estimated); Last update posted 2020-07-09 (Actual); Status verified 2018-02

CONDITIONS: Heart Failure; Ventricular Dysfunction; Cardiomyopathies; Heart Diseases; Cardiovascular Diseases
Keywords: Cardiac Resynchronization Therapy; cardiac pacing; electrical stimulation; bi-ventricular pacing
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction; Cardiomyopathies; Heart Diseases; Cardiovascular Diseases | interventions — Mutagenesis, Insertional

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Implant (Experimental): Implant of the WiCS-LV system
  Interventions: Device: WiCS-LV system

INTERVENTIONS:
Device: WiCS-LV system — Wireless cardiac stimulator implant to pace the left ventricle for CRT Transvascular endocardial implantation of wireless pacing Electrode and subcutaneous implantation of Implantable Pulse Generator
  Other Names: Implant

SUMMARY:
The study is intended to demonstrate the safe implant of small receiver-electrodes into the endocardial surface of the left ventricle and to demonstrate its utility in providing cardiac resynchronization therapy in heart failure patients.

DETAILED DESCRIPTION:
Eligible patients will undergo an acoustic window assessment using transthoracic echocardiography. Patients with adequate acoustic windows will undergo implantation of the WiCS-LV system.

Patients will undergo evaluations pre-hospital discharge, and at one month, 3 months, and 6 months post implantation. Extended follow-up will be obtained via a registry at 1, 2, 3, 4, and 5 years post implantation.

ELIGIBILITY:
Inclusion Criteria:

Patients with standard indications for CRT based upon the most recent ESC/EHRA guidelines AND meeting criteria for one of these two categories:

1. Patients with previously implanted pacemakers or ICD's and meeting standard indications for CRT but in whom standard CRT is not advisable due to known high risk - referred to as "upgrades". Justifications for not using standard CRT must be documented in a CRF.
2. Patients in whom coronary sinus lead implantation or attempted implantation for CRT has failed to provide demonstrable therapy benefit - referred to as "untreated"

Exclusion Criteria:

1. Inability to comply with the study follow-up or other study requirements
2. History of chronic alcohol/drug abuse and currently using alcohol/drugs
3. Non-ambulatory (or unstable) NYHA class 4
4. Contraindication to heparin
5. Contraindication to both chronic anticoagulants and antiplatelet agents
6. Triple anticoagulation therapy (warfarin, clopidogrel, ASA, and other agents)
7. Thrombocytopenia (platelet count <150,000)
8. Contraindication to iodinated contrast agents
9. Intracardiac thrombus by transesophageal echocardiography
10. Age less than 18 years or greater than 75
11. Attempted IPG implant within 3 days
12. Life expectancy of less than 12 months
13. Chronic hemodialysis
14. Stage 4 or 5 renal dysfunction defined as GFR <30
15. Grade 4 mitral valve regurgitation
16. Myocardial infarction within one month
17. Major cardiac surgery within one month
18. History of a pericardial effusion in prior procedures
19. Female of childbearing potential, pregnant, or breastfeeding (a pregnancy test will be obtained where applicable)
20. Non-cardiac implanted electrical stimulation therapy devices

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-07; Primary Completion 2015-08 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Number of patients with device-related adverse events as a measure of safety | 24 hour peri-operative and one month
  Device-related adverse events are those in which the WiCS-LV system is directly or indirectly responsible.
Number of patients with procedure-related adverse events as a measure of safety | 24 hour perioperative and one month
  Procedure-related adverse events are those which occur during the WiCS-LV system implant procedure.
Bi-ventricular pacing capture | one month
  Bi-ventricular pacing capture documented on 12-lead EKG

SECONDARY OUTCOMES:
Number of patients with device-related adverse events as a measure of safety | 6 months
  Device-related adverse events are those in which the WiCS-LV system is directly or indirectly responsible.
Number of patients with serious adverse events as a measure of safety | 6 months
Bi-ventricular pacing capture | 6 months
  Bi-ventricular pacing capture documented on 12-lead EKG
Clinical composite score | 6 months
  Composite of all cause mortality, heart failure hospitalization, NYHA class, and patient global assessment
Change in echocardiographic indices | 6 months
  change in left-ventricular end-systolic volume, left ventricular end-diastolic volume, and ejection fraction

CONTACTS AND LOCATIONS:
Locations (2):
- Na Homolce Hospital, Prague, Czechia
- Aalborg University Hospital, Aalborg, Denmark

REFERENCES:
- [Derived] Reddy VY, Miller MA, Neuzil P, Sogaard P, Butter C, Seifert M, Delnoy PP, van Erven L, Schalji M, Boersma LVA, Riahi S. Cardiac Resynchronization Therapy With Wireless Left Ventricular Endocardial Pacing: The SELECT-LV Study. J Am Coll Cardiol. 2017 May 2;69(17):2119-2129. doi: 10.1016/j.jacc.2017.02.059. PMID 28449772